CLINICAL TRIAL: NCT04316221
Title: The Effects ofComplementary Feeding of Eggs on Infant Developmentand Growth in Guatemala: The Saqmolo Study
Brief Title: Effects of Complementary Feeding of Eggs on Infant Development and Growth in Guatemala: The Saqmolo Study
Acronym: Saqmolo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academy of Nutrition and Dietetics (Other)
Collaborators: Wuqu' Kawoq, Maya Health Alliance (Other); Think Healthy Group, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AcademyND
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Growth; Development; Delayed
Keywords: Eggs; nutrition; growth stunting; infant development
MeSH Terms: interventions — Eggs; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial involving children ages ~6 to 12 months from communities in central Guatemala within Wuqu' Kawoq's catchment area individually randomized to either the intervention or control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The standard of nutrition care in Guatemala includes the following clinical care, as determined to be necessary by the MHA medical and nutrition teams: frequent growth monitoring, general nutrition education, parasite treatment, and multiple micronutrient supplementation.
  Interventions: Other: Standar of care
- Intervention (Experimental): The intervention group will receive an intervention to promote daily egg consumption for a six month period, in addition to the local standard of nutrition care. Specifically, intervention group participants will be provided with enough eggs for the infant to consume one egg, daily, for six months, and also with education on preparation and consumption of eggs.
  Interventions: Dietary Supplement: Eggs plus standard of care

INTERVENTIONS:
Dietary Supplement: Eggs plus standard of care — Eggs will be secured locally and delivered to families weekly.
  Arms: Intervention
Other: Standar of care — frequent growth monitoring, general nutrition education, parasite treatment, and multiple micronutrient supplementation.
  Arms: Control

SUMMARY:
The specific aims of this study are:

In a randomized controlled trial, the investigators will evaluate the impact of daily egg consumption during the complementary feeding period in addition to the local standard of nutrition care (i.e., intervention group), compared to the local standard of nutrition care alone (i.e., control group) on the following outcomes, in infants that are ~6-month old at baseline:

1. Child development, as measured by global development scores (primary outcome)
2. Growth, as measured by anthropometrics (secondary outcome)
3. Diet quality, as measured by the World Health Organization infant and young child feeding indicators (secondary outcome)

Hypothesis: The investigators hypothesize that daily consumption of eggs during the complementary feeding period, in addition to the local standard of nutrition care, will improve child development, growth, and diet quality compared to the local standard of care alone.

DETAILED DESCRIPTION:
Background: Approximately 150 million children, or roughly one-quarter of children worldwide, experience stunting (low height-for-age), while 20% are underweight.1 World-wide, undernutrition is estimated to be responsible for 2.2 million deaths and 21% of Disability-Adjusted Life Years (DALYs) in children less than 5 years of age. 1 The recent United Nations Sustainable Development Goals call for reducing stunting and wasting in children <5 years by 40%, which would affect 90 million children worldwide 1.

The global attention to stunting is based on the premise that any intervention aimed at improving linear growth may subsequently lead to improvements in the correlates of stunting 2. In children, stunting is consistently associated with poor developmental outcomes3. However, optimal interventions to concurrently address stunting and child development still need to be identified3-9.

In Guatemala, stunting is a serious public health problem10,11. The overall prevalence of stunting in children under 5 years of age in Guatemala is close to 50% and is even higher (close to 70%) for indigenous children12. The majority of indigenous families in Guatemala live on less than $2 (USD) per day and have inadequate access to health and nutrition services.

Wuqu' Kawoq-Maya Health Alliance (MHA) (http://www.wuqukawoq.org) is a non-governmental organization, located in Tecpán, Guatemala, working with vulnerable indigenous communities to provide culturally and linguistically appropriate healthcare services. MHA is currently collaborating with the Academy of Nutrition and Dietetics/UNM on projects to address malnutrition in rural Guatemala.

This study will specifically focus on evaluating the impact of regular egg consumption from about 6-12 months of age, in addition to the local standard of nutrition care, as an intervention to improve development, growth and diet quality in Mayan children. Eggs are a rich source of nutrients important to child growth and development: essential fatty acids, choline, vitamins A, and B12, and bioavailable iron, zinc and iodine13. Individual components of eggs may be associated with improved cognitive development in healthy populations, as recently reviewed by Wallace14. Eggs are culturally acceptable as part of the typical Mayan diet, are generally more affordable than other animal-source foods and are relatively simple to store and prepare15. A recent study found that egg consumption (1 egg/d for 6 months) reduced stunting in mixed-indigenous rural Andean children in Ecuador by 47% (HR: 0.53; 95% CI: 0.38-0.88);16 however, child cognitive development was not assessed in this small intervention study. This study will address a gap in understanding the impact of egg consumption, combined with other common interventions to address undernutrition in low- and middle-income settings, on both child development and growth.

Study Design: This is a randomized controlled trial involving children ages ~6 to 12 months from communities in central Guatemala within Wuqu' Kawoq's catchment area (departments of Chimaltenango, Sololá, Sacatepéquez, Suchitepéquez) individually randomized to either the intervention or control group.

* The control group will receive the local standard of nutrition care only. The standard of nutrition care in Guatemala includes the following clinical care, as determined to be necessary by the MHA medical and nutrition teams: frequent growth monitoring, general nutrition education, parasite treatment, and multiple micronutrient supplementation.
* The intervention group will receive an intervention to promote daily egg consumption for a six month period, in addition to the local standard of nutrition care. Specifically, intervention group participants will be provided with enough eggs for the infant to consume one egg, daily, for six months, and also with education on preparation and consumption of eggs.

Subjects and Timeline: The study will enroll 1200 infants into two study groups: intervention (n=600 children) and control (n=600 children). The study is powered to detect a difference in effect size of 0.15 for growth, assuming a 20% attrition rate over the course of the six month study. The investigators used a smaller effect size than found in previous relevant literature, because the control group in those studies did not also receive the clinical care that is part of standard of nutrition care in Guatemala, as will be the case in this study.

This study will use a rolling recruitment approach. Approximately 40 infants per month will be enrolled into each study group. The investigators anticipate 15 months of rolling recruitment, with final subjects finishing the study at ~21 months after beginning recruitment. The expected total duration of the study, including data analysis and dissemination, is approximately 3 years from the date of IRB approval.

Individual participants and their caregivers will have approximately 10-12 hours of contact with the research team over about 6 months:

* Study enrollment (visits to recruit, assess eligibility, and complete the informed consent process) is anticipated to take ~total 2 hours.
* The primary study data collection time points will be at 0 months (baseline) and 6 months (end of standard of care/egg intervention). It is anticipated that each of these study data collection visits will last approximately 1-2 hours (~total 2-4 hours).
* All participants will have six ~60 minute visits with MHA field staff (~total 6 hours). At those visits, all participants will receive the nutrition standard of care and be screened for development of an egg allergy. The intervention group will also receive eggs and egg related education, and answer brief questions about adherence.

Research Setting: The study will be conducted with communities in Wuqu' Kawoq's catchment area (departments of Chimaltenango, Sololá, Sacatepéquez, Suchitepéquez) in central Guatemala. The primary language spoken in this area is Kaqchikel. MHA has been providing primary care and nutrition services in this area for over a decade and collaborates closely with Ministry of Health staff and multiple other non-governmental organizations in the region.

All recruitment, enrollment and study-related procedures will be conducted in the homes of the subjects. All study procedures will be conducted by MHA staff. The study will be locally overseen and approved by MHA's IRB.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are 6.0-9.0 months of age at baseline
* At least one caregiver willing to provide oral informed consent
* Planned residence in the study area for approximately the next 18 months
* Singleton birth

Exclusion Criteria:

* Infants with moderate to severe acute malnutrition (weight-for-length z-score < -2)
* Infants with severe anemia (Hgb <7 g/dL per WHO guidelines, with adjustments for altitude as necessary)
* Infants with a chronic medical condition that affects growth (e.g., congenital heart disease, genetic condition) as determined by the MHA staff physician
* Infants whose caregivers have cognitive or other impairments that prevent them from being able to provide informed consent or to reliably provide information required for the developmental assessments
* Infants with a known egg allergy
* Infants with recalcitrant, moderate-to-severe atopic dermatitis
* Infants with a history of anaphylaxis or serious allergic reaction to any substance requiring emergency medical care
* Concurrent participation in any other clinical trial

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver Reported Child Development Instruments (CREDI) | 6 months
  The long form CREDI uses caregiver report and captures five domains: motor, language, cognition, social-emotional, and mental health. The CREDI is designed specifically to measure normal development within populations and has been tested in high, middle and low income countries The CREDI included a Guatemalan sample in the validation
Guide for Monitoring Child Development (GMCD) | 6 months
  The GMCD has been used in low- and middle-income countries in children ages 0-24 months and focuses on seven areas: expressive language, receptive language, fine motor, gross motor, relating, play, and self-help.

SECONDARY OUTCOMES:
changes in infant hemoglobin | 6 months
  Point-of-care hemoglobin will be assessed using a capillary blood sample obtained from the infant's heel or finger and a HemoCue® Hb201+ promo (HemoCue AB, Angelholm, Sweden).
weight-for-age | 6 months
  weight as appropriate for chronological age. Weight will be monitored using a hanging Salter scale to the nearest 0.1 kg.
length-for-age | 6 months
  Infant length will be measured using a portable stadiometer to the nearest 1 mm.
Head circumference | 6 months
  Head circumference will be measured using non-stretchy measuring tape to the nearest 1 mm.
Infant diet quality | 6 months
  Infant diet quality will be measured using the World Health Organization Infant and Young Child Feeding indicators questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Wuqu' Kawoq/Maya Health Alliance, Tecpán Guatemala, Departamento de Chimaltenango, Guatemala

IPD SHARING:
Plan to Share IPD: No